CLINICAL TRIAL: NCT01149889
Title: An Open-label, Crossover Study on Major Depressive Disorder Using Transcranial Direct Current Stimulation
Brief Title: Transcranial Direct Current Stimulation to Treat Major Depressive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Andre Brunoni, P.I., Research Associate, University of Sao Paulo
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: USP-HU-002
Record Dates: First submitted 2010-06-22; First posted 2010-06-24 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- active stimulation (Experimental): In active stimulation, the anode is placed over the left dorsolateral prefrontal cortex and the cathode is placed over the right prefrontal cortex. They are located five centimeters ventrally of the primary motor area, which are located five centimeters laterally of the central point of the scalp (which is located on the intersection of the sagittal and median curves). The device will deliver a charge of 2mA for 30 minutes.
  Interventions: Procedure: transcranial direct current stimulation

INTERVENTIONS:
Procedure: transcranial direct current stimulation — Transcranial direct current stimulation will be applied at 2mA, 30 minutes/day, for 10 weekdays consecutively

SUMMARY:
The investigators purpose is to offer active Transcranial Direct Current Stimulation (tDCS) in patients of the investigators previous study who received either placebo or sertraline and have not responded.

ELIGIBILITY:
Inclusion criteria:

Patients from a previous study (ID:USP-HU-001) who:

* received sertraline and did not respond.
* received placebo and did not respond.

Exclusion criteria:

Patients from a previous study who:

* received active tDCS.
* responded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Treatment Response | Week 1
  Response is defined as MADRS <=12 or less than 50% of baseline MADRS (Montgomery Asberg depression rating score).
Treatment response | Week 2
  Response defined as above.

CONTACTS AND LOCATIONS:
Overall Officials: Andre R Brunoni, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil